CLINICAL TRIAL: NCT06497933
Title: Exhaustive French National Online Registry of Atrial Fibrillation Ablation Procedures Using the Pentaspline Pulsed Field Ablation Catheter
Brief Title: Exhaustive French National Registry of AF Ablation Using Pentaspline Pulsed Field Ablation Catheter
Acronym: FRANCE-PFA
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/0259/OB
Record Dates: First submitted 2024-07-04; First posted 2024-07-12 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Atrial Fibrillation
Keywords: Pulsed field ablation; registry
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Paroxysmal atrial fibrillation patients: patients with paroxysmal atrial fibrillation undergoing first time catheter ablation using the pentaspline PFA catheter
  Interventions: Procedure: Atrial fibrillation ablation
- Persistent atrial fibrillation patients: patients with persistent atrial fibrillation undergoing first time catheter ablation using the pentaspline PFA catheter
  Interventions: Procedure: Atrial fibrillation ablation
- Long-standing persistent atrial fibrillation patients: patients with long-standing persistent atrial fibrillation undergoing first time catheter ablation using the pentaspline PFA catheter
  Interventions: Procedure: Atrial fibrillation ablation

INTERVENTIONS:
Procedure: Atrial fibrillation ablation — Pulmonary veins isolation potentially associated with other atrial lesions, performed with the pentaspline PFA catheter
  Other Names: Pulsed field ablation procedure using the Faradrive catheter (Boston Scientific)

SUMMARY:
Pulsed field ablation (PFA) is a nonthermal ablative modality using a strong electrical field created around a dedicated catheter to produce pores in the cellular membrane. As the amount of energy required to produce electroporation is highly tissue dependent, the atrial myocardium can be specifically targeted while sparing adjacent tissues. This new ablation modality could increase the safety of pulmonary vein isolation (PVI) procedures compared to PVI using thermal energies. The investigators aim to provide the first exhaustive Nationwide registry using the pentaspline PFA catheter to treat atrial fibrillation patients.

DETAILED DESCRIPTION:
This is a multicenter observational research project, that prospectively included patients undergoing a first time atrial fibrillation ablation using the Farapulse technology (Boston Scientific) since the start of this technology in France.

All patients treated with the Farapulse technology for atrial fibrillation in France from March 2021 to February 29th of 2024 will be included in the registry. The number of participating centers is 33.

A one-year and 2-year follow-up will be performed according to the standard practices of the different centers. The study duration will be 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Patients who received catheter ablation for paroxysmal AF, persistent AF, or long-standing persistent AF.

Exclusion Criteria:

* Previous left atrial ablation.
* Patient's opposition to participating in this registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent for the first time an atrial fibrillation ablation procedure, with pulmonary veins isolation performed with the pentaspline PFA catheter in France will be included in the registry
Sampling Method: Non-Probability Sample
Enrollment: 5223 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
long-term efficacy (AA) | within 1-year period post-procedure
  freedom from all types of atrial arrhythmia recurrences
very long-term efficacy (AA) | Within 2 years period post-procedure
  freedom from all types of atrial arrhythmia recurrences

SECONDARY OUTCOMES:
long term efficacy (AF) | within 1-year period post-procedure
  freedom from atrial fibrillation recurrences
very long-term efficacy (AF) | Within 2 years period post-procedure
  freedom from atrial fibrillation recurrences
Safety outcomes | within 1-month post-procedure
  the composite of major adverse events, including esophageal complications, symptomatic PV stenosis, cardiac tamponade requiring intervention, stroke or systemic thromboembolism, persistent phrenic nerve injury, vascular access complications requiring surgery, coronary artery spasm, and death

CONTACTS AND LOCATIONS:
Overall Officials: Frederic ANSELME, MD, PhD, Principal Investigator — University Hospital, Rouen
Locations (1):
- University Hospital of Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chaumont C, Laredo M, Thomas O, Maury P, Massoulie G, Defaye P, Boveda S, Marijon E, Escande W, Roux A, Raczka F, Guyomar Y, Jais P, Ollitrault P, Granier M, Fareh S, Marchand H, Pierre B, Abbey S, Noel A, Da Costa A, Extramiana F, Cesari O, Champ-Rigot L, Khoueiry Z, Villemin T, Traulle S, Treguer F, Bader H, Deharo JC, Degand B, Guy-Moyat B, Klug D, Gandjbakhch E, Zhao A, Beneyto M, Eschalier R, Venier S, Combes S, Lepillier A, Mielczarek M, Clementy N, Menet A, Sacher F, De Chillou C, Anselme F. Countrywide introduction of pulsed field ablation for the treatment of atrial fibrillation: Acute results from the FRANCE-PFA registry. Heart Rhythm O2. 2025 Apr 25;6(7):911-919. doi: 10.1016/j.hroo.2025.04.005. eCollection 2025 Jul. PMID 40734736